CLINICAL TRIAL: NCT00521625
Title: Epidemiologic Multicenter Study on Mechanical Ventilation Management in Children With Acute Lung Injury - Phase 1 PALIVE 1 (for Pediatric Acute Lung Injury Mechanical VEntilation Strategies)
Brief Title: Epidemiologic Multicenter Study on Mechanical Ventilation Management in Children With Acute Lung Injury
Acronym: PALIVE1
Status: Completed | Type: Observational
Sponsor: St. Justine's Hospital (Other)
Other Study IDs: PALIVE1
Record Dates: First submitted 2007-08-24; First posted 2007-08-28 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Acute Lung Injury; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
PALIVE 1 is an observational multicenter study on mechanical ventilation strategies used in children with an acute lung injury (ALI). The objective of the study is to describe mechanical ventilation strategies in children with an ALI. Our hypothesis is that daily clinical practice is heterogenous among pediatric intensivists as few pediatric data exists on optimal mechanical ventilation strategies in this group of patients. Furthermore, different strategies may affect patient outcome.

DETAILED DESCRIPTION:
INTRODUCTION Few pediatric data exists on the ventilation mode and parameters that would provide the greatest benefit with the least risk to an individual pediatric patient with Acute Lung Injury (ALI). Current expert opinion is that it is reasonable to follow adult recommendations and to adapt clinical management in children according to adult data. In the absence of consensus and established guidelines for mechanical ventilation in children with ALI, we believe that the daily clinical practice in pediatric intensive care units is subject to great variations according to the experience, comfort and knowledge of the attending intensivist.

METHODS Objective: Describe invasive and non-invasive mechanical ventilation in pediatric cases of ALI.

Hypothesis: There is an important variability in the observed practice pattern of mechanical ventilation in pediatric cases of ALI.

Design: An international cross-sectional epidemiologic study in Pediatric Intensive Care Units on the observed practice pattern of invasive and non-invasive mechanical ventilation in children with ALI.

Setting: Pediatric Intensive Care Units in Canada, United States, Europe.

Patients: Patients less than 18 years old on invasive or non-invasive mechanical ventilation with a diagnosis of ALI on the day of the study.

Measurements: Demographic data on included patients; their underlying chronic disease and acute disease leading to non-invasive mechanical ventilation or intubation and mechanical ventilation; data on mechanical ventilation mode and parameters, vital signs, lab results, radiographic findings, treatments, complications of mechanical ventilation will be recorded every 6 hours for 24 hours. A web based case report form will be developed.

Sample size: We plan to conduct the study on isolated days at least one month apart until we reach 200 patients with ALI, to include at least 10 patients on high frequency ventilation. We estimate that with 5 days of study in 70 centers we should reach this number.

FUTURE CONSIDERATIONS We believe this study will provide important data on the actual mechanical ventilation strategies in pediatric patients with ALI. The next step will be to conduct a prospective international study on mechanical ventilation strategies and to follow patients prospectively during the whole course of their mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Child on invasive mechanical ventilation administered through an endotracheal tube or a tracheostomy tube, or on non-invasive mechanical ventilation administered through a nasal or facial mask or a nasal canula or helmet at 9 a.m. on the day of the study.
* Presence of ALI as estimated by the attending physician:

  1. Onset of hypoxemia was acute
  2. Bilateral infiltrates on chest X-Ray
  3. No clinical evidence of congestive heart failure
  4. Sustained hypoxemia defined as:

PaO2(mmHg)/FiO2 ratio ≤ 300 or PaO2(kPa)/FiO2 ≤ 40

If no arterial canula or no arterial blood gas:

SpO2/FiO2 ≤ 320 with SpO2 < 0.98 (10)

Exclusion Criteria:

* Post conceptional age < 42 weeks
* Age > 18 years
* Non-corrected cyanotic congenital heart disease or evidence of extra-pulmonary right to left shunt
* Withdrawal/withholding of care
* Brain death
* No consent, if required
* Patient on ECMO
* Already included in this study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2007-06; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Jouvet, MD, Principal Investigator — St. Justine's Hospital
Locations (58):
- United States (20):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital at Oakland, Oakland, California
  - The Children's Hospital, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Miami Children's Hospital, Miami, Florida
  - Children's Memorial Hospital, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Kentucky Children's Hospital, Lexington, Kentucky
  - UMAss Memorial Medical Center, Worchester, Massachusetts
  - Children's Mercy Hospital, Kansas City, Missouri
  - Children's Hospital, Omaha, Nebraska
  - Nebraska Medical Center, Omaha, Nebraska
  - Darmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - New York Presbyterian Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - The Children's hospital Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Austin, Austin, Texas
  - Texas Childrens Hospital, Houston, Texas
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Austria (2):
  - Akademisches Lehrkrankenhaus, Feldkirch
  - Medical University of Vienna, Vienna
- Belgium (2):
  - Paola Childrens Hospital, Antwerp
  - Cliniques universitaires Saint-Luc, Brussels
- Canada (8):
  - Hôpital SteJustine, Montreal, Quebec
  - Montreal Children' Hospital, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Stollery Children's Hospital, Edmonton
  - McMaster Children's Hospital, Hamilton
  - Children's Hospital of Western Ontario, London
  - Centre Hospitalier Universitaire de Quebec, Québec
  - BC Children's Hospital, Vancouver
- France (5):
  - CHU Lille, Lille
  - CHU Nantes, Nantes
  - Hôpital Robert-Debré, Paris
  - Necker, Paris
  - CHU Pontchaillou, Rennes
- Germany (5):
  - University Clinic Frankfurt, Frankfurt
  - Universitätsklinikum Mannheim, Mannheim
  - Kinderzentrum im Klinikum Nürnberg, Nuremberg
  - Children's Hospital StAugustin, Sankt Augustin
  - University Children's Hospital, Tuebringen
- Italy (3):
  - Ospedali riuniti di Bergamo, Bergamo
  - Padua University Hospital, Padua
  - Azienda Ospedaliera di Verona, Verona
- The Wilhelmina Children's Hospital, Utrecht, Netherlands
- Spain (7):
  - Hospital Sant Joan de Déu-Hospital Clinic, Barcelona
  - Cruces Hospital, Bilbao
  - General University Hospital Gregorio Marañón, Madrid
  - Hospital Universitario Central de Asturias, Oveido
  - Hospital universitario de Salamanca, Salamanca
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Infantil La Fe, Valencia
- Sweden (2):
  - The Queen Silvia Children's Hospital, Gothenburg
  - Astrid Lindgren Children's Hospital, Stockholm
- Switzerland (2):
  - Children's Hospital, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
- Bristol Children's Hospital, Bristol, United Kingdom

REFERENCES:
- See also: Web site for the study's data collection — http://palive1.crc.chus.qc.ca/